CLINICAL TRIAL: NCT03641248
Title: Study to Establish the Bioavailability and Pharmacokinetic Measures of H. Procumbens Extract in Humans
Brief Title: Bioavailability and Pharmacokinetic Measures of H. Procumbens Extract
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Recruitment was not possible due to COVID19.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, William Folk, Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2010425; US NIH Grant 7R21AT009086 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2018-08-16; First posted 2018-08-21 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Harpagophytum extract LI 174

STUDY DESIGN:
Intervention Model Description: Pharmacokinetic
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enteric coated Devil's Claw (Experimental): H. procumbens 100 mg in enteric coated capsules
  Interventions: Drug: Enteric coated Devil's Claw
- Non-enteric coated Devil's Claw (Active Comparator): H. procumbens 100 mg in non-enteric coated capsules
  Interventions: Drug: Non-enteric coated Devil's Claw

INTERVENTIONS:
Drug: Enteric coated Devil's Claw — Enteric coated capsules containing Devil's Claw extract with 100mg harpagoside
  Other Names: Harpagophytum procumbens
  Arms: Enteric coated Devil's Claw
Drug: Non-enteric coated Devil's Claw — Non-enteric coated capsules containing Devil's Claw extract with 100mg harpagoside
  Other Names: Harpagophytum procumbens
  Arms: Non-enteric coated Devil's Claw

SUMMARY:
Study will define the bioavailability and short term pharmacokinetics of the principal secondary metabolites of a aqueous-ethanolic extract of H. procumbens in non-enteric and enteric capsules.

DETAILED DESCRIPTION:
The study(n = 12) will use a one-dose design to measure bioavailability and pharmacokinetic properties of an aqueous extract of H. procumbens containing 100mg harpagoside. Plasma levels of harpagoside, harpagide, verbascoside, and 8-p-coumarylharpagide will be measured for 24 hours with blood collections taken at timed intervals.

ELIGIBILITY:
Inclusion Criteria:- adult (at least 18 years of age);

* diagnosed with knee osteoarthritis (OA) ;
* body mass index (BMI) of less than 40;
* willing to use only the study product, and Tramadol or Tylenol as a rescue pain medication over the course of their participation in the study;
* willing and able to monitor blood glucose levels if diabetic;
* willing to abstain from caffeine-containing drinks and food before coming into a study visit;
* able to read and understand English and have the cognitive capacity to give consent;
* willing to abstain from use of the following during participation in the study: prescription and over-the-counter non-steroidal anti-inflammatory medications, (e.g., aspirin, ibuprofen, Advil, Motrin, Nuprin, Naproxen, etc.); any dietary supplements (St. John's Wort, etc.); and, grapefruit and/or products containing it.

Exclusion Criteria:- cardiovascular disease, previous myocardial infarction, stent, coronary artery bypass graft (CABG), arrhythmia, high or low blood pressure;

* recurrent stomach upset, or gastric or duodenal ulcers;
* gallstones or gall bladder disease (cholelithiasis);
* liver or kidney disease;
* alcohol use of more than two drinks per day on a regular basis;
* Coumadin or anti-platelet drug use;
* at risk for respiratory depression, history of seizures, or taking drugs that reduce the seizure threshold or may increase the risk for development of serotonin syndrome;
* pregnant or breast feeding, or intention to become pregnant during the study;
* pronounced allergies, or known allergy to study product or corn starch (placebo);
* have had an injection to treat OA within the past three months;
* currently taking NSAIDs, unless they are willing to stop for a 1-week wash-out period;
* currently on a selective serotonin reuptake inhibitor (SSRI) but are poorly stabilized, or have evidence of suicidal ideation and/or suicide attempts in the past year; and,
* reported use during the 7 days prior to study drug administration of: prescription and over-the-counter medications (e.g., NSAIDs), and any dietary supplements; grapefruit and/or its products; and, St. John's Wort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Maximal concentration level of Devil's Claw metabolites, Cmax (ng/ml) | 0.5 hour, 1 hour, 2 hours, 2.5 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 9 hours, 10 hours, 12 hours
  Blood will be drawn at predefined intervals following administration of one dose of study drug
Time to reach Cmax (h) | 0 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours
  Blood will be drawn at predefined intervals following administration of one dose of study drug
Determination of terminal half-life of Devil's Claw, t 1/2 (h) | 0 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours
  Blood will be drawn at predefined intervals following administration of one dose of study drug

SECONDARY OUTCOMES:
Change in plasma levels of harpagoside | 24 hours after dose of Devil's Claw
  Blood will be drawn for Devil's Claws metabolites at Visit 2
Change in plasma levels of harpagide | 24 hours after dose of Devil's Claw
  Blood will be drawn for Devil's Claws metabolites at Visit 2
Change in plasma levels of verbascoside | 24 hours after dose of Devil's Claw
  Blood will be drawn for Devil's Claws metabolites at Visit 2
Change in levels of 8-p-coumarylharpagide | 24 hours after dose of Devil's Claw
  Blood will be drawn for Devil's Claws metabolites at Visit 2

CONTACTS AND LOCATIONS:
Overall Officials: William Folk, PhD, Principal Investigator — Univ of Missouri
Locations (1):
- Univ of Missouri Health Care Center, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT03641248/Prot_ICF_000.pdf